CLINICAL TRIAL: NCT01878695
Title: Pilot Study of Anti-oxidant Supplementation With N-Acetyl Cysteine in Stage 0/I Breast Cancer
Acronym: NAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12D.396; JT 2312 (Other: JeffTrial Number)
Record Dates: First submitted 2013-06-11; First posted 2013-06-17 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Stage 0/1 Breast Cancer; Post Biopsy; Pre-surgery
Keywords: Integrative Medicine; Breast Cancer; Stage 0; Stage 1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV and oral n-acetylcysteine (Experimental): 50-150mg/kg of n-acetylcysteine intravenously once a week for at least two weeks.
  600mg n-acetylcysteine orally twice daily except on day of infusion
  Interventions: Drug: IV/oral n-acetylcysteine

INTERVENTIONS:
Drug: IV/oral n-acetylcysteine

SUMMARY:
NAC is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine. It is a common over-the-counter supplement and also is available as an injectable pharmaceutical that protects the liver in cases of acetaminophen overdose. In the exercise physiology literature, both oral and injectable NAC have been shown to reduce fatigue and improve recovery from exertion which has interesting implications for exploring cancer-related fatigue.

In terms of cancer cell biology, reactive oxygen species (ROS) may play an important role in the development and progression of breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Demographic • Females ≥18 years of age

Disease related

* Stage 0/I breast cancer by biopsy (patients may be consented and screened with suspected breast cancer, but no treatment will occur until cancer is confirmed by their biopsy).
* Awaiting surgery which will consist of either lumpectomy or mastectomy.
* ECOG performance status 0-1

Laboratory

* Laboratory values that would not prevent the patient from receiving treatment as determined by the PI or study oncologist
* Serum creatinine ≤2.0 mg/dL
* Serum bilirubin ≤2.0 X ULN
* Serum HgB ≥8.0 mg/dL

General

* Competent to comprehend, sign, and date an IRB-approved informed consent form
* Female subjects of childbearing potential have a negative pregnancy test

Exclusion Criteria:

* Disease Related

  * History or known presence of metastases
  * History of another primary cancer, except:
* Curatively treated cervical carcinoma in situ, or
* Curatively resected non-melanomatous skin cancer, or
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≤ 3 years prior to enrollment

  * Other concurrent anticancer chemotherapy within 4 weeks as determined by the PI
  * Any co-morbid disease that would increase risk of toxicity as determined by PI

Medications/Treatments

* Subjects requiring chronic use of immunosuppressive agents (eg, methotrexate, cyclosporine, corticosteroids)
* Recent infection requiring a course of systemic anti-infectives that was completed ≤ 14 days prior to enrollment (exception can be made at the judgment of the PI for oral treatment of an uncomplicated urinary tract infection ([UTI])

General

* History of any medical or psychiatric condition or addictive disorder, or laboratory abnormality that, in the opinion of the PI, may increase the risks associated with study participation or study drug administration or may interfere with the conduct of the study or interpretation of study requirements
* History of bronchospasm or severe asthma as determined by the PI
* Subject unwilling or unable to comply with study requirements
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* Documented history of alcohol, cocaine or intravenous drug abuse ≤ 6 months of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07-26 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2-4 weeks
  To assess the feasibility of evaluating the effect of n-acetylcysteine on tumor cell metabolism by assessing the changes in expression of caveolin -1 and MCT4 in cancer associated fibroblasts in pre and post therapy breast tissue treated with NAC.

SECONDARY OUTCOMES:
Safety | 2-4 weeks
  To confirm the safety of combined oral and IV NAC in patients with breast cancer. This will be evaluated by the number of participants with adeverse events and Grade 3/4 toxicities according to CTCAE v3.0
2. To access the changes in HIF-1 alpha and p65 subunit of NFB in tumor stroma in pre and post therapy breast tissue treated with NAC | 2-4 weeks
  To access the changes in HIF-1 alpha and p65 subunit of NFB in tumor stroma in pre and post therapy breast tissue treated with NAC
To evaluate potential effects of NAC on quality of life and fatigue | 2-4 weeks
  To evaluate potential effects of NAC on quality of life and fatigue using the FACT-G, Brief Fatigue Inventory, and PROMIS quality assessment instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Monti, MD, MBA, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Jefferson Myrna Brind Center for Integrative Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/